CLINICAL TRIAL: NCT07027202
Title: Early Preventive Left Ventricle Unloading After VA-ECMO for Refractory Cardiogenic Shock
Acronym: EULODIA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: APHP240927; IDRCB Number (Other: 2024-A02655-42)
Record Dates: First submitted 2025-05-07; First posted 2025-06-18 (Actual); Last update posted 2025-06-18 (Actual); Status verified 2025-05

CONDITIONS: Cardiogenic Shock Acute
Keywords: ECMO; BPIA; Cardiogenic shock acute

STUDY DESIGN:
Intervention Model Description: Multicenter, prospective, randomized, comparative open trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Early Left Ventricle unloading arm (Experimental): An Intraortic balloon pump will be systematically inserted as soon as possible, within 12 hours post-randomization.
  * A pulmonary artery catheter (PAC) will enable hemodynamic monitoring of cardiac filling pressures, cardiac output and pulmonary artery pressures.
  * Doppler Echocardiography will be performed at least daily to monitor LV ejection, LV dimension, appearance of LV blood stagnation, aortic time-velocity integral (VTI) and aortic valve opening.
  * Escalation to a microaxial LV venting pump, central ECMO or atrial septostomy will be possible and discussed by the Shock team (as suggested by international recommendations) in case of
  * Overt cardiogenic pulmonary edema requiring invasive mechanical ventilation
  * Persisting more than 6 hours despite IABP support and optimization of patient's management (titration of ECMO blood flow, inotropes, non-invasive mechanical ventilation with PEEP, diuretics or hemofiltration).
  Interventions: Procedure: Early Left Ventricle unloading
- Standard management of VA-ECMO cardiogenic shock patients. (No Intervention): A pulmonary artery catheter will enable hemodynamic monitoring of cardiac filling pressures, cardiac output, and pulmonary artery pressures. - Doppler Echocardiography will be performed at least daily to monitor LV ejection, LV dimension, appearance of LV blood stagnation, aortic VTI and aortic valve opening. - Optimization of patient's management in case of signs of cardiogenic pulmonary edema occurring under VA-ECMO (titration of ECMO blood flow, inotropes, non-invasive ventilation mechanical ventilation with PEEP, diuretics or hemofiltration). - LV unloading (IABP, microaxial LV venting pump, central ECMO or atrial septostomy) (as suggested by international recommendations) discussed by the Shock team in case of overt cardiogenic pulmonary edema persisting more than 6 hours despite the aforementioned measure and the recourse to invasive mechanical ventilation AND o PCWP >20 mmHg OR o Aortic valve opening less than 50% of electric systole and VTI < 4cm

INTERVENTIONS:
Procedure: Early Left Ventricle unloading — An Intraortic balloon pump will be systematically inserted as soon as possible, within 12 hours post-randomization.
  * A pulmonary artery catheter (PAC) will enable hemodynamic monitoring of cardiac filling pressures, cardiac output and pulmonary artery pressures.
  * Doppler Echocardiography will be performed at least daily to monitor LV ejection, LV dimension, appearance of LV blood stagnation, aortic time-velocity integral (VTI) and aortic valve opening.
  * Escalation to a microaxial LV venting pump, central ECMO or atrial septostomy will be possible and discussed by the Shock team (as suggested by international recommendations) in case of
  * Overt cardiogenic pulmonary edema requiring invasive mechanical ventilation
  * Persisting more than 6 hours despite IABP support and optimization of patient's management (titration of ECMO blood flow, inotropes, non-invasive mechanical ventilation with PEEP, diuretics or hemofiltration).
  Arms: Early Left Ventricle unloading arm

SUMMARY:
Venoarterial extracorporeal membrane oxygenation (VA-ECMO) is increasingly being used worldwide to treat severe cardiogenic shock. The survival rate of these patients has increased in the last decade, reaching 45-50% for patients with acute myocardial infarction (AMI), the most frequent indication of the technique, 50-60% for patients with end-stage dilated cardiomyopathy bridged to heart transplantation or long-term left ventricle assist device (LVAD) surgery, 60-70% for fulminant myocarditis, while it remains lower for post-cardiotomy cardiogenic shock (25-35%) and after cardiac arrest (20-40%). However, peripherally inserted VA-ECMO increases left ventricular (LV) afterload, that may lead to poorer clinical outcomes by fostering left ventricular distension, blood stagnation, aortic valve closure, all of which increasing pulmonary congestion and the need for mechanical ventilation and compromising myocardial recovery whenever it is possible, or delaying a bridge to a heart transplantation or long-term left ventricle assist device (LVAD) surgery for patients with end-stage cardiac dysfunction. Several methods have been proposed to reduce afterload after VA-ECMO, including the use of an intra-aortic balloon pump (IABP), balloon atrial septostomy, transseptal left atrial cannula insertion, and use of the left-sided Impella device (Abiomed, Danvers, MA, USA). The clinical benefits of left ventricular unloading have been suggested by many retrospective case-control studies, including a study by our group that showed that associating an IABP with peripheral VA-ECMO was independently associated with a lower frequency of hydrostatic pulmonary edema under ECMO and more days off mechanical ventilation. More recently, unloading the left ventricle with an IABP was associated with the best survival rate and security profile as compared to no unloading or unloading with a microaxial pump in 12,734 VA-ECMO patients included in the Extracorporeal Life Support Organization registry. It should also be mentioned that another large registry study showed that the greatest benefit of LV unloading under ECMO was observed with early versus delayed insertion of the unloading device. Lastly, the EARLY-UNLOAD randomized trial in which a transseptal left atrial cannula was used for LV unloading yielded negative results. However, it is important to note that 50% of control patients were rapidly transitioned to LV unloading, thereby compromising the opportunity to demonstrate a mortality benefit. It was also underpowered for the primary outcome of D30 mortality since it included only 116 patients As a result, the recourse to systematic early LV unloading remains highly heterogeneous in clinical practice. For example, , while IABP was EULODIA - Protocol, version 1.0 dated 24/01/2025 Page 6 sur 54 This document is the property of DRCI/AP-HP. All reproduction is strictly prohibited.

Version no. 4.0 of 31/05/2019 associated to ECMO in >70% of the cases in our series of AMI CS patients, only 5.8% of the patients included in the ECMO arm of the recent ECLS-Shock trial received an unloading device, which may have contributed to the neutral result of the study and the only randomized trial to date was underpowered and flawed by a very high rate of early cross-over. Indeed, there is large heterogeneity in current clinical practice, where decisions on whether to add an additional mechanical unloading device during VA-ECMO support vary widely.

Therefore, a new and adequately powered trial comparing systematic early left ventricular unloading to a conventional approach, with rescue left ventricular unloading only in case of clear and urgent indication, i.e. if overt hydrostatic cardiogenic pulmonary edema occurs, is urgently needed. The EULODIA trial is designed to test the hypothesis that early preventive left ventricle unloading with an IABP improves clinical outcomes as compared to conventional care with delayed curative unloading in patients under VA-ECMO for refractory cardiogenic shock.

ELIGIBILITY:
Inclusion Criteria:

1. Patient on peripheral femoro-femoral VA ECMO for severe Cardiogenic shock for ≤24h
2. Initiation of LV unloading possible within 12 hours after randomization.
3. Consent obtained from a close relative or surrogate. Should such a person be absent, eligible patients will be randomized according to the specifications of emergency consent and the patient will be asked to give his/her consent for the continuation of the trial when his/her condition will allow.
4. Social security registration (AME excluded)

Exclusion Criteria:

1. Age <18 years
2. Pregnancy
3. Onset of VA-ECMO >24 h
4. Overt pulmonary edema despite optimization of patient's management (titration of ECMO blood flow, inotropes, non-invasive mechanical ventilation with PEEP, diuretics or hemofiltration) requiring urgent LV unloading
5. ECMO for massive pulmonary embolism or primary RV failure
6. ECMO after heart transplant
7. ECMO after LVAD surgery
8. Resuscitation >30 minutes before ECMO (cumulative low-flow time), except if the patient has fully recover consciousness at the time of randomization.
9. ECMO for refractory cardiac arrest (E-CPR)
10. Grade 3-4 aortic regurgitation
11. Mechanical complication of acute myocardial infarction (massive mitral regurgitation, pericardium drainage required, septal ventricular defect)
12. Patient moribund on the day of randomization
13. Cerebral deficit with fixed dilated pupils or Irreversible neurological pathology
14. Other severe concomitant disease with limited life expectancy <1 year
15. Patient has a durable ventricular assist device, an IABP or another temporary mechanical circulatory support (other than ECMO) prior to enrollment.
16. Severe peripheral artery disease or previous aortic or ilio-femoral surgery precluding IABP or IMPELLA insertion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 298 (Estimated)
Dates: Start 2025-06 (Estimated); Primary Completion 2027-07 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
Composite hierarchical outcome assessed at day 30, composed of three components: 1)All-cause mortality, 2)unloading device or strategy related complication 3) time off temporary mechanical circulatory support (tMCS) or invasive mechanical ventilation ( | Day 30
  o Each subject is compared to every other subject and assigned one number resulting from each pair-wise comparison (win +1; lose-1; tie=0) based on whom fared better. Since mortality outcome is clinically more important, mortality takes precedence over complications and days off IMV/tMCS at day 30. If one patient survived at day 30 and the other did not, scores of +1 and -1 will be assigned, respectively. If both patients survived, the assigned score will depend on the second component: if one patient had a complication and the other did not, a score of -1 and +1 will be assigned, respectively. If both patients survived without complication, the assigned score will depend on which patient had more time off t-MCS/IMV: the patient with more time off will receive a score of +1, and the other -1. For each patient, scores for all pairwise comparisons will be summed, resulting in a cumulative score which will be the primary endpoint of the study

SECONDARY OUTCOMES:
Bleeding (BARC 3 or more) | Day 30
Infection at any MCS insertion site treated by antibiotics | Day 30
Critical limb ischemia (leading to fasciotomy, surgical or endovascular intervention, MCS withdrawal). | Day 30
Stroke (ischemic or hemorrhagic) | Day 30
Any specific complication associated with intraventricular microvascular pump (aortic or mitral valve lesion, severe hemolysis) or atrial septostomy (tamponade, cardiac perforation). | Day 30
All-cause mortality | Day 60
Duration of ECMO support | Day 60
Bridge to durable ventricular assist device (left ventricular assist device type Heartmate3 or a total artificial heart) or heart transplantation | Day 60
Durations of ICU stay | Day 60
Number of days of invasive mechanical ventilation | Day 30
Number of days of renal replacement therapy | Day 30
Number of days alive without organ failure(s) | From randomization to day 30
Number of ventilator-associated pneumonia treated with antibiotics | From randomization to Day 60
Durations of hospitalization | Day 60
Durations of ICU stay | Between inclusion and Day 30
Durations of hospitalization | Between inclusion and Day 30
Major complication specifically related to the unloading device (IABP, microaxial IMPELLA pump) or strategy (atrial septostomy) - Bleeding (BARC 3 or more) | Between inclusion and Day 30
All cause mortality | Day 30
Number of days of ECMO support and days free of ECMO support | Day 30
Delay to overt pulmonary edema (defined by pulmonary capillary wedge pressure (PCWP) >20 mmHg and bilateral infiltrates on Chest X-ray) indicating escalation to an unloading device (IABP, microaxial LV venting pump or atrial septostomy for control group | Day 30
Rate of bridge to durable ventricular assist device or heart transplantation | Day 30
Total number of packed red blood cells and platelet transfused | Day 30
Left ventricular function assessed with Doppler echocardiography for alive patients only | Day 30

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume LEBRETON, MD, Study Director — Assistance Publique Hôpitaux de Paris - Pitié Salpêtrière Hospital; Adrien BOUGLE, MD, Study Director — Assistance Publique Hôpitaux de Paris - Pitié Salpêtrière Hospital

IPD SHARING:
Plan to Share IPD: Yes
The procedures carried out with the French data privacy authority (CNIL, Commission nationale de l'informatique et des libertés) do not provide for the transmission of the database, nor do the information and consent documents signed by the patients.
  Consultation by the editorial board or interested researchers of individual participant data that underlie the results reported in the article after deidentification may nevertheless be considered, subject to prior determination of the terms and conditions of such consultation and in respect for compliance with the applicable regulations.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Beginning 3 months and ending 3 years following article publication. Requests out of these time frame can also be submitted to the sponsor
Access Criteria: Researchers who provide a methodologically sound proposal